CLINICAL TRIAL: NCT02395289
Title: The Efficacy of Cognitive-Based Compassion Training for Enhancing Immune Restoration and Psychological Adaptation in Individuals Living With HIV Disease
Brief Title: Cognitive-Based Compassion Training (CBCT) for People Living With HIV (PLHIV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Mehul Tejani, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00075221
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: Cognitive-Based Compassion Training (CBCT); HIV-related clinical outcomes; Stress and stress-related psychological adjustment; Stress-related inflammatory biomarkers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Based Compassion Training (CBCT) (Experimental): HIV-1 positive subjects on antiretroviral therapy (ART) will be randomized to receive an 8-week program of Cognitive-Based Compassion Training (CBCT).
  Interventions: Behavioral: Cognitive-Based Compassion Training (CBCT)
- Health Discussion Control (Active Comparator): HIV-1 positive subjects on antiretroviral therapy (ART) will be randomized to attend a health discussion group for 8 weeks.
  Interventions: Behavioral: Health discussion

INTERVENTIONS:
Behavioral: Cognitive-Based Compassion Training (CBCT) — Cognitive-Based Compassion Training (CBCT) is composed of secular, didactic instruction and meditation practices. CBCT includes the meditative practices of developing one-pointed concentration and mindfulness. CBCT will be one class per week, 2 hours each, for 8 weeks, for a total of 16 hours during the study. Each meditation class will include a didactic and discussion session that will describe the meditative technique introduced during the week and a practice meditation session. The training protocol is highly iterative and techniques introduced early in training are practiced daily. All participants will be asked to meditate approximately 30 minutes a day "at home" and will be given a meditation diary to record amount of time spent meditating per week.
  Arms: Cognitive-Based Compassion Training (CBCT)
Behavioral: Health discussion — Health discussion therapy is one class per week, 2 hours each, for 8 weeks. Each class will use interactive teaching methods to present the health material in an engaging and relevant manner. Representative weekly topics that will be covered include healthy diet, the role of exercise in emotional health, and the importance of sleep and relaxation. It is important to note that the material presented in the health discussion group, although intended to be beneficial to participants, does not include a contemplative component and is not iterative in nature.
  Arms: Health Discussion Control

SUMMARY:
The purpose of the study is to examine the effects of cognitive-based compassion training (CBCT), a meditative practice based on Buddhist teachings, on long term emotional well-being and immune system improvement with people living with Human Immunodeficiency Virus (PLHIV).

DETAILED DESCRIPTION:
The proposed study will investigate the efficacy of cognitive-based compassion training (CBCT), a contemplative technique based on the Tibetan Buddhist tradition of compassion meditation, for enhancing immune restoration and psychological resilience in people living with HIV-1 (PLHIV). Psychosocial stress has been associated with increased circulating concentrations of key inflammatory biomarkers. The patients with HIV must cope with the physical impact of HIV disease itself, the often complex treatment regimens and side effects of combination antiretroviral therapy (ART), illness-associated psychological and existential dilemmas, changes in social roles and lifestyle patterns relative to illness progression, social stigma, and financial and material resource concerns. This study aims to determine if engagement with CBCT is associated with reduced circulating concentrations of stress-related inflammatory biomarkers, improves HIV-related clinical outcomes and decreases stress in PLHIV.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects living with HIV-1 infection who have been on continuous ART for a minimum of 12 months and:

   * are followed longitudinally for their HIV healthcare at the Infectious Disease Program
   * meet criteria for immunological non-responsiveness as defined by adherence to ART and cluster of differentiation 4 (CD4) count <350 cells/μL despite complete virologic suppression (> 2 plasma HIV viral load (pVL) below the limit of detection including the most recent pVL prior to enrollment).
2. Ability to give informed consent.
3. Score at least 1 standard deviation above socioeconomic status (SES)-matched general population norms on Perceived Stress Scale (PSS)

Exclusion Criteria:

1. History of psychosis
2. HIV-related neurocognitive decline
3. Substance abuse within the last year
4. Documented history of cirrhosis or a total bilirubin ≥ 2.0 mg/dL
5. Known or possible pregnancy or attempting to become pregnant
6. BMI below 17 or above 30
7. Age < 18
8. Bipolar disorder
9. Bleeding disorders such as thrombocytopenia or significant gastrointestinal bleeding within the past year
10. Continuous ART for < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentration of circulating inflammatory biomarker interleukin-6 (IL-6) | screening, 8 weeks
  The plasma concentrations of IL-6 will be assessed using commercial enzyme-linked immunoassay (ELISA) kits.
Change in plasma concentration of circulating inflammatory biomarker soluble cluster of differentiation 14 (sCD14) | screening, 8 weeks
  The plasma concentrations of sCD14 will be assessed using commercial enzyme-linked immunoassay (ELISA) kits.

SECONDARY OUTCOMES:
Change in scores on the Perceived Stress Scale (PSS) | Screening, 8 weeks
  The PSS is a 10-item scale that provides a general index of perceived psychological stress as this relates to a sense that one's life is experienced as unpredictable, uncontrollable, and overloaded. The subjects are asked to indicate how often they felt or thought a certain way and to score their responses on a scale from 0 to 4, where 0= Never and 4=Very Often. PSS is measured on a scale of 0 to 40, with higher scores reflecting greater perceived stress.
Change in scores on the General Well-Being (GWB) Schedule Scale | Screening, 8 weeks
  The GWB is an 18-item self-report scale designed to measure subjective psychological well-being and distress. It includes six subscales (anxiety, depression, positive well-being, self-control, vitality, general health) and also yields an overall well-being score. The response format used a 6-grade Likert scale and the range of scores will be normalized from 0 to 100. The higher the score, the better the well-being of the participant.
Change in scores on the Illness Cognition Questionnaire (ICQ) | Screening, 8 weeks
  This ICQ is an 18-item self-report measure used to assess changes in illness appraisal. It includes three subscales that evaluate specific dimensions of illness cognitions. Each of the three scales (helplessness, acceptance and benefits) consists of 6 items that are rated according to a 4-point Likert scale to the extent of agreement (0= not at all, 1=somewhat, 2= to a large extent, 3= completely), producing a total score ranging from 0 to 72, with a higher score being indicative of more illness appraisal.
Change in scores on the World Assumptions Scale (WAS) | Screening, 8 weeks
  The WAS is a 32-item self-report instrument that measures core personal beliefs. Subscales tap specific core belief domains, including: benevolence of the impersonal world, benevolence of people, justice, controllability of life events, self-worth, self-controllability, and personal luck. Each of these scales consist of items that are rated according to a 6-point Likert-type scale bounded by 1 (strongly disagree) and 6 (strongly agree). The higher the score is indicative to a stronger belief.
Change in scores on the Life Regard Index - Revised (LRI-R). | Screening, 8 weeks
  The LRI-R is a 28-item scale that provides an index of global personal meaning. It includes two subscales: framework (assesses one's sense of having a frame of reference from which to appraise one's life and goals), and fulfillment (evaluates the degree to which one perceives that life goals are being realized). Both of these scales consist of items that are rated according to a 3-point Likert scale (1= I agree, 2= I have no opinion and 3= I disagree) and scores on both subscales range between 14 and 42, for a total range of 28 and 84. In case of the framework subscale, a higher score indicates a higher degree of positive beliefs and goals. In case of the fulfillment subscale, a higher score indicates that persons see themselves in the process of fulfilling their beliefs and goals.
Change in scores on the Rosenberg self-esteem scale | Screening, 8 weeks
  The Rosenberg Self-esteem scale is a 10-item scale that provides a self-report index of self-esteem. Each item is rated according to a 4-point Likert scale with scores ranging from strongly agree to strongly disagree. The scale ranges from 0-30, with 30 indicating the highest score possible. Total sum scores between 15 and 25 are within normal range; with scores below 15 suggest low self-esteem.
Change in scores on the Berger HIV Stigma Scale | Screening, 8 weeks
  The Berger HIV Stigma Scale is a 13-item self-report measure that evaluates perceptions of HIV stigma across three subscale domains, including distancing (concerns about avoidance by others), blaming (feelings of blame from others and internal shame relative to HIV), and discrimination (concerns about inequitable treatment because of HIV). Each item is rated according to a 4-point Likert scale with scores ranging from bounded by 1 (strongly disagree) and 4 (strongly agree). Endorsement of stigmatizing views yielded a higher score.
Change in serum levels of C-reactive protein (CRP) | Screening, 8 weeks
  The serum concentration of CRP will be assessed using commercial enzyme-linked immunoassay (ELISA) kits.
Acceptance of Cognitive-Based Compassion Training (CBCT), measured by participant satisfaction | 8 weeks
  Acceptance of the CBCT will be measured by positive responses on a participant satisfaction survey, developed specifically for the study, which will be conducted at the completion of the 8-week program.

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Tejani, MD, Principal Investigator — Emory University
Locations (1):
- Grady Hospital - Ponce De Leon Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Titanji BK, Tejani M, Farber EW, Mehta CC, Pace TW, Meagley K, Gavegnano C, Harrison T, Kokubun CW, Negi SD, Schinazi RF, Marconi VC. Cognitively Based Compassion Training for HIV Immune Nonresponders-An Attention-Placebo Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2022 Mar 1;89(3):340-348. doi: 10.1097/QAI.0000000000002874. PMID 34879006